CLINICAL TRIAL: NCT06401109
Title: Evaluating the Safety and Efficacy of the AquaPass System a Renal-independent Fluid Removal System in ADHF Patients Suffering From Fluid Overload. a European Registry
Brief Title: Naturally Controlled Decongestion Using Renal Independent System in ADHF Patients, a European Registry
Acronym: REFORM-HF II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AquaPass Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQP-CLP-044
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Chronic Heart Failure; Fluid Overload; Acute Decompensated Heart Failure; Edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AquaPass (Experimental): Patients hospitalized with chronic heart failure symptoms and fluid overload will be treated in two phases:
  Phase 1: 'In Hospital' Phase: Patients will be enrolled in the study when admitted to the hospital with fluid overload.
  Use of the AquaPass system will be performed in the hospital, alongside diuretic therapy.
  Phase 2: 'At Home' Phase: Upon the investigator's decision at discharge, the patients will be enrolled in this phase of the study, and will receive AquaPass treatment sessions at their home.
  Interventions: Device: AquaPass

INTERVENTIONS:
Device: AquaPass — The AquaPass system works by activating the body's natural sweating mechanism to remove excess fluid from the interstitial compartment. This process is achieved by wearing a garment that creates optimal microclimate conditions around the skin.
  The system is controlled by a portable unit that delivers warm air to the wearable component while ensuring patient safety.

SUMMARY:
The AquaPass is a non-invasive, renal-intended system designed to enhance fluid transfer through the skin, by increasing sweat rate, to treat fluid overload in heart failure patients.

This study will further evaluate the safety, efficacy, and usability of the AquaPass system in the hospital and home settings.

DETAILED DESCRIPTION:
The AquaPass system is non-invasive and functions independently of the renal system, targeting the direct removal of fluids directly from the interstitial compartment through the skin, by activating the eccrine sweat glands.

The patient wears a component that is connected to a control unit, which induces warm air to create a controlled environment around the skin, stimulating sweat production. The sweat evaporates instantly, ensuring that the patient remains dry and comfortable.

In this study, the investigators would like to further investigate the efficacy of the system, when used in hospital settings in patients hospitalized for decompensated heart failure and fluid overload, and to continue the treatment in their homes, immediately after the hospitalization, for another 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject that was hospitalized with fluid overload and a history of chronic heart failure and CKD stages 1-4
* Subject has composite congestion score ≥3.
* Baseline systolic blood pressure at rest of ≥100mmHg.
* Subject is capable of meeting the following study requirements:
* For patients with BMI <30 kg/m2: baseline NT-pro BNP>1,600 pg/ml
* For patients with BMI >30 kg/m2: baseline NT-pro BNP >800 pg/ml
* For patients with rate-controlled persistent or permanent AF: NT-pro BNP >2,400 pg/ml.
* Subject successfully completes 2-4 hours of run-in acclimation session
* Minimal sweat rate in the last hour of run-in acclimatization of 130gr/hours

Exclusion Criteria:

* Subject is enrolled to another clinical investigation that might interfere with this study.
* Baseline systolic blood pressure <100 mm Hg
* Subject considered to be in the acute worsening of the heart failure: Requiring ventilation, mechanical support or is clinically unstable requiring pressors, deterioration triggered by arrythmia, infection or other medical condition unrelated to fluid overload.
* Subject has any known lower body skin problems (open wounds, ulcers)
* Subject with severe peripheral arterial disease
* Subject is pregnant or planning to become pregnant within the study period, or lactating mothers.
* End-stage renal disease (eGFR<15 ml/min/1.73 m2) or requiring dialysis.
* Inability or unwillingness to comply with the study requirements.
* History of heart transplant or actively listed for heart transplant or Left Ventricular Assist Device (LVAD).
* Implanted left ventricular assist device or implant anticipated <3 months.
* Malignancy or other noncardiac condition limiting life expectancy to <12 months.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Average Sweat Rate Per Hour per patient | 30 days
  An average sweat rate of 150 ml/hr per patient at hospital and at home
Incidence of device- and procedure-related side-effects | 30 days
  Incidences of system and treatment-related AEs and SAEs including symptomatic changes in vital signs

SECONDARY OUTCOMES:
Incidence of worsening renal function | 30 days
  Incidence of worsening renal function, measured as an increase of Creatinine levels by >0.5mg/dL
Fluid Overload Related Hospitalizations | 30 days
  Hospitalization or ED visit for decompensated heart failure
Changes in congestion score | 30 days
  to evaluate the effect of the AquaPass treatment on congestion score
Changes in Diuretics Dose | 30 days
  Documentation of changes in diuretics administration to assess safety and potential benefits with system use.
Change of quality of life | 30 days
  Assessment of the quality of life using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The minimal score is zero '0' and the highest is '100' when higher scores represent a better outcome for the patient.
Changes in NT-ProBNP levels | 30 days
  Changes in NT-ProBNP levels to demonstrate the system's safety and clinical performance
Change in body weight | 30 days
  To evaluate the effectiveness of the AquaPass System. During the study patients will weighed before and after each treatment. The weight before the first treatment and the weight after the last treatment will be used to assess the treatment performance

IPD SHARING:
Plan to Share IPD: Undecided